CLINICAL TRIAL: NCT00458003
Title: Phenylephrine Versus Ephedrine to Treat Spinal Anesthesia-Induced Hypotension in Preeclamptic Patients During Cesarean Delivery
Brief Title: Phenylephrine in Spinal Anesthesia in Preeclamptic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Walega, Research Vice Chair Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524-31
Record Dates: First submitted 2007-04-04; First posted 2007-04-09 (Estimated); Results first posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Preeclampsia; Hypotension
Keywords: Preeclampsia; Spinal Anesthesia; Hypotension; Cesarean Delivery; Phenylephrine; Ephedrine
MeSH Terms: conditions — Pre-Eclampsia; Hypotension | interventions — Ephedrine; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phenylephrine (Experimental): Subject will receive a phenylephrine infusion to prevent and to treat hypotension associated with spinal anesthesia
  Interventions: Drug: Phenylephrine
- Ephedrine (Active Comparator): Subject will receive an ephedrine infusion to prevent and to treat hypotension associated with spinal anesthesia
  Interventions: Drug: Ephedrine

INTERVENTIONS:
Drug: Ephedrine — Ephedrine concentration: 8 mg/mL. The infusion will be initiated immediately after completion of the spinal injection at a rate of 1 mL/min and continued for a minimum of 2 min after which the infusion will be stopped, continued or increased based on the SBP each minute. After each SBP measurement the infusion will be stopped if SBP > 80% baseline, and the infusion will be continued or restarted if the SBP is approximately equal to 80% baseline. The infusion will be increased by 1 mL/min if the SBP < 80% baseline. Each time there is hypotension the patient will receive a 1 mL IV bolus of the study solution and the infusion will be increased by 1 mL/min until delivery.
  Arms: Ephedrine
Drug: Phenylephrine — Phenylephrine concentration: 100 mcg/mL. The infusion will be initiated immediately after completion of the spinal injection at a rate of 1 mL/min and continued for a minimum of 2 min after which the infusion will be stopped, continued or increased based on the SBP each minute. After each SBP measurement the infusion will be stopped if SBP > 80% baseline, and the infusion will be continued or restarted if the SBP is approximately equal to 80% baseline. The infusion will be increased by 1 mL/min if the SBP < 80% baseline. Each time there is hypotension the patient will receive a 1 mL IV bolus of the study solution and the infusion will be increased by 1 mL/min until delivery.
  Arms: Phenylephrine

SUMMARY:
Hypotension remains a common clinical problem after induction of spinal anesthesia for cesarean delivery. Maternal hypotension has been associated with considerable morbidity (maternal nausea and vomiting and fetal/neonatal acidemia). Traditionally, ephedrine has been the vasopressor of choice because of concerns about phenylephrine's potential adverse effect on uterine blood flow. This practice was based on animal studies which showed that ephedrine maintained cardiac output and uterine blood flow, while direct acting vasoconstrictors, e.g., phenylephrine, decreased uteroplacental perfusion. However, several recent studies have demonstrated that phenylephrine has similar efficacy to ephedrine for preventing and treating hypotension and may be associated with a lower incidence of fetal acidosis. All of these studies have been performed in healthy patients undergoing elective cesarean delivery.

Preeclampsia complicates 5-6% of all pregnancies and is a significant contributor to maternal and fetal morbidity and mortality. Many preeclamptic patients require cesarean delivery of the infant. These patients often have uteroplacental insufficiency. Given the potential for significant hypotension after spinal anesthesia and its effect on an already compromised fetus, prevention of (relative) hypotension in preeclamptic patients is important. Spinal anesthesia in preeclamptic patients has been shown to have no adverse neonatal outcomes as compared to epidural anesthesia when hypotension is treated adequately. Due to problems related to management of the difficult airway and coagulopathy, both of which are more common in preeclamptic women, spinal anesthesia may be the preferred regional anesthesia technique. Recent studies have demonstrated that preeclamptic patients may experience less hypotension after spinal anesthesia than their healthy counterparts. To our knowledge, phenylephrine for the treatment of spinal anesthesia-induced hypotension has not been studied in women with preeclampsia. The aim of our study is to compare intravenous infusion regimens of phenylephrine versus ephedrine for the treatment of spinal anesthesia induced hypotension in preeclamptic patients undergoing cesarean delivery. The primary outcome variable is umbilical artery pH.

DETAILED DESCRIPTION:
The study will be approved by the Northwestern University Institutional Review Board. Eligible women admitted to the Labor and Delivery Unit of Prentice Women's Hospital will be approached for study participation immediately after the routine preanesthetic evaluation. This usually occurs shortly after admission to the Labor and Delivery Unit. Women who agree to participate will give written, informed consent at this time.

Preparation and initiation of spinal anesthesia will proceed according to routine practice at our institution. A 16-gauge IV catheter will be inserted under local anesthesia in the pre-operative labor and delivery suite. An IV infusion of lactated Ringer's solution will be started at a minimal rate to maintain vein patency. Patients will be premedicated with metoclopramide 10 mg and ranitidine 50 mg IV at least 30 minutes prior to procedure for aspiration prophylaxis. Patients will be allowed to rest undisturbed for several minutes in the left lateral tilt position, during which heart rate (HR) and systolic blood pressure (SBP) will be taken every 1-2 minutes for at least 3 measurements. Baseline HR and SBP will be the mean of these three recordings.

The subjects will be randomized according to a computer-generated randomization table to one of two groups: Group 1 will receive a phenylephrine infusion and Group 2 will receive an ephedrine infusion. All study medications will be prepared by an investigator not involved in the care of the patient or collection of data. Both the anesthesiologist managing the patient's anesthetic, as well as the patient, will be blinded to the study medication.

Upon arrival to the operating room, 30 mL of 0.3 M sodium citrate will be given orally and standard monitoring will performed, including non-invasive BP, electrocardiography and pulse oximetry. Oxygen will be given at 3 liter per minute by nasal cannula. Fetal heart rate will be monitored by external cardiotocography until the time of surgical preparation. 500 mL of lactated Ringer's solution will be given as a bolus concurrently with the start of the spinal anesthesia procedure. Spinal anesthesia will be induced with patients in the sitting position. After sterile skin preparation and draping, the skin will be infiltrated with lidocaine, a 25 gauge Whitacre needle will be inserted at the L3-L4 vertebral interspace (± one vertebral interspace) and bupivacaine 0.75%, 1.6 mL (12 mg), fentanyl 15 μg and morphine 150 μg will be injected intrathecally. Patients will be immediately placed supine with left uterine displacement. SBP will be measured every 1 minute beginning 1 minute after spinal injection for 10 minutes, then every 2.5 minutes for the remainder of the procedure. Patients' hemodynamic data will be recorded throughout the procedure and printed at the end of the surgery. Five minutes after spinal injection, the sensory level of anesthesia will be assessed by loss of pinprick discrimination using von Frey hairs. If the patient fails to obtain at least a T6 sensory level of anesthesia, that patient will be withdrawn from the study. Preincision antibiotics, magnesium sulfate and uterotonic agents will be administered intraoperatively per routine practice.

An unblinded investigator will prepare solutions of phenylephrine 100 μg per mL and ephedrine 8000 μg per mL (potency phenylephrine:ephedrine 80:111). The investigator will place 20 mL of the study medication into a syringe which will be given to the managing anesthesiologist for infusion via a syringe pump. The infusion will be attached to the IV cannula at the most distal. The infusion will be initiated immediately after completion of the spinal injection at a rate of 1 mL per minute and continued for a minimum of two minutes after which the infusion will either be stopped, continued or increased based on the SBP measurement each minute. The goal will be to maintain SBP ≥ 80% baseline, but not > 160 mmHg. After each measurement of SBP, the infusion will be stopped if the SBP is greater than 80% baseline SBP, and the infusion will be continued or restarted if the SBP is approximately equal to 80% baseline SBP.12 The infusion will be increased by 1 mL per minute if the SBP measurement is less than 80% baseline. For the purpose of this study, we will define hypotension as a decrease in SBP to < 80% of baseline.13 Each time there is a SBP measurement demonstrating hypotension as defined above, the patient will receive a 1 mL IV bolus of the study solution via the infusion pump and the infusion will be increased by 1 mL per minute. The infusion and bolus protocol will be continued until delivery, after which further management will be at the discretion of the managing anesthesiologist to maintain SBP. If the baseline SBP > 160 mmHg, the infusion will not be started until the SBP decreases to 160 mmHg. Infusion management will then proceed as described above.

The total volumes of the study solutions given by infusion and bolus up to the time delivery will be recorded. Bradycardia (defined as HR < 60 bpm) associated with an SBP equal or greater to baseline SBP will be treated by stopping the study solution and bradycardia associated with SBP < 80% baseline will be treated with atropine intravenously. Hypotension unresponsive to study medication will be treated with epinephrine (10 μg/mL) intravenous boluses (1 mL) until correction of hypotension. Nausea or vomiting not associated with hypotension will be treated with ondansetron 4 mg IV.

After delivery, oxytocin 10-20 IU will be given by slow IV infusion per routine. The infant's 1 and 5 minute Apgar scores will be assessed by the nurse or pediatrician blinded to patient group. The results of routine umbilical cord blood gas analysis will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA PS II - III women
* 18 years old and older
* scheduled for cesarean delivery (no trial of labor)
* eligible for spinal anesthesia
* diagnosis of preeclampsia

Exclusion Criteria:

* patients with failed trial of labor
* preexisting hypertension
* body mass index (BMI) ≥ 40 kg/m2
* resting heart rate < 60 bpm
* progression to eclampsia, > twin gestation
* known fetal anomalies
* contraindications to spinal anesthesia
* emergency procedure or refusal of consent
* failure to achieve a T6 level of anesthesia
* conversion to general anesthesia

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2006-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Walega, M.D., Study Chair — Northwestern University
Locations (2):
- United States (2):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Northwestern University, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rout CC, Rocke DA. Prevention of hypotension following spinal anesthesia for cesarean section. Int Anesthesiol Clin. 1994 Spring;32(2):117-35. No abstract available. PMID 8063445
- [Background] Ayorinde BT, Buczkowski P, Brown J, Shah J, Buggy DJ. Evaluation of pre-emptive intramuscular phenylephrine and ephedrine for reduction of spinal anaesthesia-induced hypotension during Caesarean section. Br J Anaesth. 2001 Mar;86(3):372-6. doi: 10.1093/bja/86.3.372. PMID 11573527
- [Background] Lee A, Ngan Kee WD, Gin T. A quantitative, systematic review of randomized controlled trials of ephedrine versus phenylephrine for the management of hypotension during spinal anesthesia for cesarean delivery. Anesth Analg. 2002 Apr;94(4):920-6, table of contents. doi: 10.1097/00000539-200204000-00028. PMID 11916798
- [Background] Cooper DW, Carpenter M, Mowbray P, Desira WR, Ryall DM, Kokri MS. Fetal and maternal effects of phenylephrine and ephedrine during spinal anesthesia for cesarean delivery. Anesthesiology. 2002 Dec;97(6):1582-90. doi: 10.1097/00000542-200212000-00034. PMID 12459688
- [Background] Ngan Kee WD, Khaw KS, Ng FF, Lee BB. Prophylactic phenylephrine infusion for preventing hypotension during spinal anesthesia for cesarean delivery. Anesth Analg. 2004 Mar;98(3):815-21, table of contents. doi: 10.1213/01.ane.0000099782.78002.30. PMID 14980943
- [Background] James PR, Nelson-Piercy C. Management of hypertension before, during, and after pregnancy. Heart. 2004 Dec;90(12):1499-504. doi: 10.1136/hrt.2004.035444. No abstract available. PMID 15547046
- [Background] Report of the National High Blood Pressure Education Program Working Group on High Blood Pressure in Pregnancy. Am J Obstet Gynecol. 2000 Jul;183(1):S1-S22. PMID 10920346
- [Background] Visalyaputra S, Rodanant O, Somboonviboon W, Tantivitayatan K, Thienthong S, Saengchote W. Spinal versus epidural anesthesia for cesarean delivery in severe preeclampsia: a prospective randomized, multicenter study. Anesth Analg. 2005 Sep;101(3):862-868. doi: 10.1213/01.ANE.0000160535.95678.34. PMID 16116005
- [Background] Aya AGM, Mangin R, Vialles N, Ferrer JM, Robert C, Ripart J, de La Coussaye JE. Patients with severe preeclampsia experience less hypotension during spinal anesthesia for elective cesarean delivery than healthy parturients: a prospective cohort comparison. Anesth Analg. 2003 Sep;97(3):867-872. doi: 10.1213/01.ANE.0000073610.23885.F2. PMID 12933418
- [Background] Aya AGM, Vialles N, Tanoubi I, Mangin R, Ferrer JM, Robert C, Ripart J, de La Coussaye JE. Spinal anesthesia-induced hypotension: a risk comparison between patients with severe preeclampsia and healthy women undergoing preterm cesarean delivery. Anesth Analg. 2005 Sep;101(3):869-875. doi: 10.1213/01.ANE.0000175229.98493.2B. PMID 16116006
- [Background] Saravanan S, Kocarev M, Wilson RC, Watkins E, Columb MO, Lyons G. Equivalent dose of ephedrine and phenylephrine in the prevention of post-spinal hypotension in Caesarean section. Br J Anaesth. 2006 Jan;96(1):95-9. doi: 10.1093/bja/aei265. Epub 2005 Nov 25. PMID 16311286
- [Background] Ngan Kee WD, Khaw KS, Ng FF. Prevention of hypotension during spinal anesthesia for cesarean delivery: an effective technique using combination phenylephrine infusion and crystalloid cohydration. Anesthesiology. 2005 Oct;103(4):744-50. doi: 10.1097/00000542-200510000-00012. PMID 16192766
- [Background] Ngan Kee WD, Khaw KS, Ng FF. Comparison of phenylephrine infusion regimens for maintaining maternal blood pressure during spinal anaesthesia for Caesarean section. Br J Anaesth. 2004 Apr;92(4):469-74. doi: 10.1093/bja/aeh088. Epub 2004 Feb 20. PMID 14977792
- [Derived] Higgins N, Fitzgerald PC, van Dyk D, Dyer RA, Rodriguez N, McCarthy RJ, Wong CA. The Effect of Prophylactic Phenylephrine and Ephedrine Infusions on Umbilical Artery Blood pH in Women With Preeclampsia Undergoing Cesarean Delivery With Spinal Anesthesia: A Randomized, Double-Blind Trial. Anesth Analg. 2018 Jun;126(6):1999-2006. doi: 10.1213/ANE.0000000000002524. PMID 28953494

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The number of women enrolled in the study.
Period: Overall Study
Arm/Group | Phenylephrine | Ephedrine
Started | 55 | 55
Completed | 54 | 54
Not Completed | 1 | 1
Not completed — Non protocol spinal anesthesia | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phenylephrine | Ephedrine | Total
Number analyzed (Participants) | 54 | 54 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 54 | 108
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 54 | 108
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 54 | 54 | 108
Estimated gestational age (weeks) [Mean (Full Range); unit: weeks] — Estimated gestational age in weeks.
  weeks | 36 [33 to 37] | 36 [34 to 37] | 36 [33 to 37]
Multiple gestation [Count of Participants; unit: Participants] — The number of participants with multiple gestation.
  Participants | 18 | 20 | 38
Preeclampsia [Count of Participants; unit: Participants] — Preeclampsia defined by the American College of Obstetricians and Gynecologist before 2013 (mild or severe).
  Participants
    Mild preeclampsia | 27 | 26 | 53
    Severe preeclampsia | 27 | 28 | 55
Number of infants delivered per group [Number; unit: number of infants] — Total number of infants per group in the study. 108 participants delivered 146 babies.
  number of infants | 72 | 74 | 146
Baseline systolic blood pressure [Median (Full Range); unit: mmHg] — The average of 3 systolic blood pressures reported as mmHg obtained before spinal anesthesia procedure.
  mmHg | 150 [139 to 162] | 146 [136 to 157] | 148 [136 to 162]
Baseline heart rate [Median (Full Range); unit: Number] — Average of 3 heart rate (beats per minute) averaged for baseline prior to the start of spinal anesthesia procedure.
  Number | 83 [75 to 94] | 85 [76 to 95] | 84 [75 to 95]
Body mass index [Median (Full Range); unit: kg/m^2] — Body mass index defined as BMI (kg/m^2).
  kg/m^2 | 31 [28 to 37] | 33 [29 to 36] | 32 [28 to 37]

OUTCOME MEASURES:

1. Primary Outcome: The Umbilical Artery pH
Description: The umbilical artery blood pH immediately after delivery. The pH scale ranges from 0 to 14. A normal pH sample from the umbilical artery ranges from pH: 7.18 - 7.38.
  The lower the pH the more acidic and the higher the pH the more basic.
Time Frame: Immediately after delivery
Population: 72 newborn blood samples in the phenylephrine group and 74 newborn blood samples were analyzed (there were multiple gestations in both groups)
Measure: Median (Standard Deviation); unit: pH
Units Other Than Participants: Newborn blood gas samples
Arm/Group | Phenylephrine | Ephedrine
Number analyzed (Participants) | 54 | 54
Number analyzed (Newborn blood gas samples) | 72 | 74
pH | 7.22 (.07) | 7.20 (.1)
Statistical Analysis 1: Comparison: Phenylephrine vs Ephedrine; Test type: Superiority; p = .38, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: The Umbilical Artery Blood Base Excess
Description: The umbilical artery blood base excess immediately after delivery. Base excess and base deficit refer to an excess or deficit, in the amount of base present in the blood.
  The value (-2 to +2 normal range) is usually reported as a concentration in units of mEq/L, with positive numbers indicating an excess of base and negative a deficit
Time Frame: Immediately after delivery
Population: 72 newborn blood samples were obtained from the phenylephrine group and 74 newborn samples were obtained from the ephedrine group ( there were multiple gestations in both groups)
Measure: Median (Full Range); unit: mEq/L
Units Other Than Participants: Newborn blood gas samples
Arm/Group | Phenylephrine | Ephedrine
Number analyzed (Participants) | 54 | 54
Number analyzed (Newborn blood gas samples) | 72 | 74
mEq/L | -2.8 [-4.6 to -2.2] | -3.4 [-5.7 to -2.0]
Statistical Analysis 1: Comparison: Phenylephrine vs Ephedrine; Test type: Superiority; p = .10, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Up to 3 hours after delivery.
Description: There were 54 women in each group (phenylephrine and ephedrine group). The women delivered 146 neonates (multiple gestations in each group) 72 neonates were delivered in the phenylephrine group and 74 neonates were delivered in the ephedrine group.
Groups:
- Phenylephrine Mothers: Subject will receive a phenylephrine infusion to prevent and to treat hypotension associated with spinal anesthesia
  Phenylephrine: Phenylephrine concentration: 100 mcg/mL. The infusion will be initiated immediately after completion of the spinal injection at a rate of 1 mL/min and continued for a minimum of 2 min after which the infusion will be stopped, continued or increased based on the SBP each minute. After each SBP measurement the infusion will be stopped if SBP > 80% baseline, and the infusion will be continued or restarted if the SBP is approximately equal to 80% baseline. The infusion will be increased by 1 mL/min if the SBP < 80% baseline. Each time there is hypotension the patient will receive a 1 mL IV bolus of the study solution and the infusion will be increased by 1 mL/min until delivery.
- Ephedrine Mothers: Subject will receive an ephedrine infusion to prevent and to treat hypotension associated with spinal anesthesia
  Ephedrine: Ephedrine concentration: 8 mg/mL. The infusion will be initiated immediately after completion of the spinal injection at a rate of 1 mL/min and continued for a minimum of 2 min after which the infusion will be stopped, continued or increased based on the SBP each minute. After each SBP measurement the infusion will be stopped if SBP > 80% baseline, and the infusion will be continued or restarted if the SBP is approximately equal to 80% baseline. The infusion will be increased by 1 mL/min if the SBP < 80% baseline. Each time there is hypotension the patient will receive a 1 mL IV bolus of the study solution and the infusion will be increased by 1 mL/min until delivery.
- Phenylepherine Infants: Infant of mother who received phenylephrine infusion to prevent and to treat hypotension associated with spinal anesthesia
  Phenylephrine: Phenylephrine concentration: 100 mcg/mL. The infusion will be initiated immediately after completion of the spinal injection at a rate of 1 mL/min and continued for a minimum of 2 min after which the infusion will be stopped, continued or increased based on the SBP each minute. After each SBP measurement the infusion will be stopped if SBP > 80% baseline, and the infusion will be continued or restarted if the SBP is approximately equal to 80% baseline. The infusion will be increased by 1 mL/min if the SBP < 80% baseline. Each time there is hypotension the patient will receive a 1 mL IV bolus of the study solution and the infusion will be increased by 1 mL/min until delivery.
- Ephedrine Infants: Infant of mothers who received an ephedrine infusion to prevent and to treat hypotension associated with spinal anesthesia
  Ephedrine: Ephedrine concentration: 8 mg/mL. The infusion will be initiated immediately after completion of the spinal injection at a rate of 1 mL/min and continued for a minimum of 2 min after which the infusion will be stopped, continued or increased based on the SBP each minute. After each SBP measurement the infusion will be stopped if SBP > 80% baseline, and the infusion will be continued or restarted if the SBP is approximately equal to 80% baseline. The infusion will be increased by 1 mL/min if the SBP < 80% baseline. Each time there is hypotension the patient will receive a 1 mL IV bolus of the study solution and the infusion will be increased by 1 mL/min until delivery.
Arm/Group | Phenylephrine Mothers | Ephedrine Mothers | Phenylepherine Infants | Ephedrine Infants
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/54 | 0/72 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54 | 27/72 | 25/74
Other Adverse Events (participants affected / at risk) | 21/54 | 28/54 | 0/72 | 0/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phenylephrine Mothers (N=54) | Ephedrine Mothers (N=54) | Phenylepherine Infants (N=72) | Ephedrine Infants (N=74)
Fetal Hypoxia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 27 (27) | 25 (25) — Fetal hypoxia as defined as a umbilical cord blood pH of 7.2. 72 infants in the phenylephrine group and 74 infants in the ephedrine group were analyzed. There were multiple gestations in each group of original participants.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phenylephrine Mothers (N=54) | Ephedrine Mothers (N=54) | Phenylepherine Infants (N=72) | Ephedrine Infants (N=74)
Reactive hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 18 (18) | 22 (22) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
We assumed that the potency of phenylephrine to ephedrine was 80:1 based on published works. Baseline BP on day of procedure may be elevated due to anxiousness. The definition of preeclampsia as defined by ACOG changed during study period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No